CLINICAL TRIAL: NCT04949009
Title: Avatrombopag in the Treatment of Primary Immune Thrombocytopenia(ITP): a Single-arm, Multi-centre, Observational Study
Brief Title: Avatrombopag in the Treatment of Primary Immune Thrombocytopenia(ITP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Proff, Shandong University
Other Study IDs: SKX-2007
Record Dates: First submitted 2021-05-13; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: Avatrombopag,Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with primary immune thrombocytopenia (ITP): Ever been diagnosed as ITP patients. The diagnostic criteria comply with the "Chinese Guidelines for the Diagnosis and Treatment of Adult Primary Immune Thrombocytopenia (2020 Edition)"
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — Avatrombopag is an orally bioavailable, small molecule thrombopoietin receptor agonist that has been developed by Dova Pharmaceuticals for the treatment of thrombocytopenic disorders.
  Other Names: Doptelet

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other well-known hospitals in China. Aims at evaluating effectiveness and safety of avatrombopag in the treatment of primary immune thrombocytopenia.

DETAILED DESCRIPTION:
The investigators are undertakingSingle-arm, multi-Centre, Observational study of 400 Patients with primary immune thrombocytopenia (ITP) from Qilu Hospital of Shandong University and other well-known hospitals in China. ITP patients will be given one tablet (20 mg) of avatrombopag daily.If the platelet count is higher than 150×10^9/L, the dose should be reduced. Prolonged dosing intervals or a combination of reduced daily dose are preferred.If the drug was taken for ≥1 week and the platelet count was still less than 30×10^9/L, the dosage should be increased. The maximum dose is 40 mg daily. Aplatelet count,AE, laboratory parameters, ECG, vital signs and other symptoms will be evaluated before and after treatment. Adverse events will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18+ years, male or female;
2. Ever been diagnosed as ITP patients. The diagnostic criteria comply with the "Chinese Guidelines for the Diagnosis and Treatment of Adult Primary Immune Thrombocytopenia (2020 Edition)"

   1. At least 2 consecutive blood tests showed a decrease in platelet count; no obvious abnormality in the morphology of blood cells by peripheral blood smear microscopy.
   2. Spleen is generally not enlarged.
   3. Bone marrow examination: the morphological characteristics of bone marrow cells in ITP patients were increased or normal megakaryocytes with maturation disorders.
   4. Other secondary thrombocytopenia must be excluded: autoimmune diseases, thyroid disease, lymphoproliferative disorders, myelodysplastic syndrome (MDS), aplastic anemia (AA), various malignant hematologic diseases, tumor infiltration, Chronic liver disease, hypersplenism, common variant immunodeficiency disease (CVID), infection, vaccination causing secondary thrombocytopenia; Thrombocytopenia due to depletion; Drug induced thrombocytopenia; Alloimmune thrombocytopenia; Thrombocytopenia during pregnancy; Congenital thrombocytopenia and pseudo-thrombocytopenia;
3. ECOG general status score ≤ 2;
4. Platelet count < 30×10^9/L；platelet count ≥< 30×10^9/L accompanied by active bleeding; If the platelet count is around 30×10^9/L and no active bleeding, a second examination must be performed to further confirm the platelet count.
5. Voluntarily signed the informed consent.
6. Any other circumstances that the investigator considers appropriate for the patient to participate in the study.

Exclusion Criteria:

1. Patients with secondary thrombocytopenia.
2. Currently receiving other TPO-RAs, rhIL-11 and rhTPO treatment, and subjects are unwilling to switch to avatrombopag treatment.
3. Patients with severe insufficiency of heart, lung, liver and kidney.
4. Pregnant or breast-feeding, or contraceptive measures cannot be taken during the trial.
5. Subjects participated in clinical studies of other investigational drugs or devices within 30 days prior to screening.
6. Having a history of psychotropic drug abuse and unable to quit or having mental disorders.
7. Having significant factors that affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.
8. Subject is allergic to avatrombopag or any of its excipients;
9. Any other circumstances that the investigator considers inappropriate for the patient to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Aged 18+ years, male or female;
  2. Ever been diagnosed as ITP patients. The diagnostic criteria comply with the "Chinese Guidelines for the Diagnosis and Treatment of Adult Primary Immune Thrombocytopenia (2020 Edition)"
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving platelet response on day 28 of treatment | on day 28 of treatment
  Percentage of participants achieving platelet response on day 28 of treatment. Platelet response rate refers to the platelet count PLT≥30×109/L and increases at least 2 times from the baseline value without bleeding in the absence of remedial therapy.

SECONDARY OUTCOMES:
Percentage of participants achieving platelet response on day 8 of treatment. | on day 8 of treatment.
  Percentage of participants achieving platelet response on day 8 of treatment. Platelet response rate refers to the platelet count PLT≥30×109/L and increases at least 2 times from the baseline value without bleeding in the absence of remedial therapy.
Percentage of participants achieving platelet response on day 14 of treatment. | on day 14 of treatment.
  Percentage of participants achieving platelet response on day 14 of treatment. Platelet response rate refers to the platelet count PLT≥30×109/L and increases at least 2 times from the baseline value without bleeding in the absence of remedial therapy.
Changes in participants' bleeding scores. | through study completion, an average of 6 months
  Thrombocytopenia bleeding scoring system is used to evaluate the changes in participants' bleeding scores.
Evaluation of adverse effects related to avatrombopag. | through study completion, an average of 6 months
  Evaluation of adverse effects related to avatrombopag including side effect,toxic reaction,post effect,anaphylactic reaction.

OTHER OUTCOMES:
Percentage of participants achieving platelet response (R) at the second month of treatment. | at the second month of treatment
  Percentage of participants achieving the platelet count PLT≥30×109/L and increases at least 2 times from the baseline value without bleeding in the absence of remedial therapy at the second month of treatment.
Participants' 6-month continuous remission rate. | 6 month of treatment
  Percentage of participants achieving 6-month continuous remission including symptoms associated with bleeding and mental symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD PhD, Principal Investigator — Shandong University Qilu Hospital
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Dlugosz-Danecka M, Zdziarska J, Jurczak W. Avatrombopag for the treatment of immune thrombocytopenia. Expert Rev Clin Immunol. 2019 Apr;15(4):327-339. doi: 10.1080/1744666X.2019.1587294. Epub 2019 Mar 8. PMID 30799645
- [Background] Shirley M. Avatrombopag: First Global Approval. Drugs. 2018 Jul;78(11):1163-1168. doi: 10.1007/s40265-018-0949-8. PMID 29995177
- [Background] Cheloff AZ, Al-Samkari H. Avatrombopag for the treatment of immune thrombocytopenia and thrombocytopenia of chronic liver disease. J Blood Med. 2019 Sep 5;10:313-321. doi: 10.2147/JBM.S191790. eCollection 2019. PMID 31565009
- [Background] Bussel JB, Kuter DJ, Aledort LM, Kessler CM, Cuker A, Pendergrass KB, Tang S, McIntosh J. A randomized trial of avatrombopag, an investigational thrombopoietin-receptor agonist, in persistent and chronic immune thrombocytopenia. Blood. 2014 Jun 19;123(25):3887-94. doi: 10.1182/blood-2013-07-514398. Epub 2014 May 6. PMID 24802775